CLINICAL TRIAL: NCT02219971
Title: Randomized, Double-blind Placebo-controlled Phase I Study to Assess Safety, Tolerance and Pharmacokinetics of a Single Intravenous Injection Kukoamine B Mesilate in Healthy Volunteers
Brief Title: Phase I Study of Kukoamine B Mesilate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Chasesun Pharmaceutical Co., LTD (Industry)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-KB101; ChiCTR-TRC-14005111 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Kukoamine B Mesilate 0.005mg/kg (Experimental): Pre-test,open study: Kukoamine B Mesilate 0.005mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.02mg/kg + Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.02mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.04mg/kg +Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.04mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.08mg/kg + Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.08mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.12mg/kg + Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.12mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.24mg/kg + Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.24mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.48mg/kg + Placebo (Experimental): Dose Escalation: Kukoamine B Mesilate 0.48mg/kg single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Placebo: single and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate

INTERVENTIONS:
Drug: Kukoamine B Mesilate — Kukoamine B Mesilate or placebo single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.

SUMMARY:
The purpose of this study is to assess safety, tolerance and pharmacokinetics of a single intravenous injection Kukoamine B Mesilate in health volunteer

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female, each sex ratio does not exceed 2/3;
* 18-45 years (including upper and lower limit), the general situation is good;
* Body mass index (BMI) in 19-28 (including upper and lower limit of the range), BW ≥ 50kg (female) and 60kg (male);
* Nearly half of the year, no child care program and agreed to take effective measures to contraception during the study period, women of childbearing age blood pregnancy test was negative;
* Subjects to fully understand the purpose, properties, method and reactions may occur of test drug trials.Voluntarily signed the informed consents, and agreed to abide by the requirements of clinical protocols.

Exclusion Criteria:

* Primary disease in important organs;
* Mental or physical disability;
* Familial hereditary disease;
* Screening supine blood pressure (after 5 minutes of rest) systolic or diastolic blood pressure greater than 90~140mmHg, beyond the scope of 50~90mmHg, Or pulse (HR) beyond 50bpm~100bpm
* Abnormal results of any clinically meaningful physical examination, vital signs, ECG or clinical laboratory;
* History of immunodeficiency diseases, including HIV antibody positive;
* Detection of antibody positive, hepatitis B surface antigen or antibody to hepatitis C / syphilis positive;
* Alcohol and drug abusers;
* Smoking and drinking are (drinking 14 units of alcohol per week: 1 unit = beer 285 ml, or liquor 25 ml, or wine 1 cup. numbers of daily smoking ≥ 5) and / or not smoking and drinking in the test period;
* Any discharge period may affect the study drug, or in the past 3 months participated in any drug clinical trials;
* Before entering the group 4 weeks using any prescription drugs before entering the group, or use of any non prescription drugs within 2 weeks (vitamins, herbal tonics, food additives), or into the group within 2 weeks before taking effect of drug metabolizing enzymes in food, such as grapefruit or grapefruit drink. Can the use of acetaminophen, but must record report in CRF;
* The last 3 months had a history of blood donation or significant blood loss (more than 400ml);
* There are drugs, the clinical significance of the history of food allergy and atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known drug to test drugs or similar drug allergy test;
* Lactating women, pregnant women or unable to take effective contraceptive measures;
* Researchers believe that the other is not suitable to take the test factors participants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2015-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events. | 7 days
  AE,physical examination,monitoring of vital signs, Laboratory examination,ECG etc.

SECONDARY OUTCOMES:
Pharmacokinetic parameters (t1/2,AUC0-inf,AUClast and Cmax;Fe0-48h(%),CLr24h) | 48h
  Blood:（Pre Test）0,20min,40min after initiation of drug administration and 0,10min,20min,30min,45min,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h,24h after the end of administration;(Formal Test) 0,20min,40min after initiation of drug administration and 0,30min,1h,2h,3h,4h,6h,8h,12h,16h,24h after the end of administration; Urine:(Pre Test) 0,0-4h,4-8h,8-12h,12-24h,24-48h after initiation of drug administration;(Formal Test) 0,0-5h,5-9h,9-13h,13-25h,25-49h after initiation of drug administration .

CONTACTS AND LOCATIONS:
Overall Officials: SHUAI CHEN, Study Director — TIAN JIN CHASE SUN PHARMACEUTICAL CO.,LTD
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu H, Zhao Q, Yuan Y, Wang Z, Wang T, Tian W, Zhong W, Jiang J, Chen S, Kong K, Jin C, Hu P. First-in-Human Safety, Tolerability, and Pharmacokinetics of Single-Dose Kukoamine B Mesylate in Healthy Subjects: A Randomized, Double-Blind, Placebo-Controlled Phase I Study. Infect Dis Ther. 2024 Feb;13(2):361-371. doi: 10.1007/s40121-024-00921-6. Epub 2024 Jan 30. PMID 38291280